CLINICAL TRIAL: NCT04592289
Title: Short-term Outcomes of Full Bowel Preparation (MBP+OA) for Rectal Resections for Cancer Versus MBP Alone
Acronym: REPCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL-3
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; bowel preparation; MBP; Oral antibiotics
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full bowel preparation (MBP+OA) (Experimental): Rifaximin 400 mg twice daily for three days prior to surgery
  Day prior to surgery:
  17.00 - 18.00 Macrogol-3350 - 100 g Sodium sulfate - 7,5 g Sodium chloride - 2,691 g Potassium chloride - 1,015 g Ascorbic acid - 4,7 g Sodium ascorbate - 5,9 g Clear fluids - 1000 ml
  18.00 - 19.00 Clear fluids 500 ml
  19.00 - 20.00 17.00 - 18.00 Macrogol-3350 - 100 g Sodium sulfate - 7,5 g Sodium chloride - 2,691 g Potassium chloride - 1,015 g Ascorbic acid - 4,7 g Sodium ascorbate - 5,9 g Clear fluids - 1000 ml
  20.00 - 21.00 Clear fluids 500 ml
  Interventions: Procedure: Full bowel preparation
- Mechanical bowel preparation only (Active Comparator): Day prior to surgery:
  17.00 - 18.00 Macrogol-3350 - 100 g Sodium sulfate - 7,5 g Sodium chloride - 2,691 g Potassium chloride - 1,015 g Ascorbic acid - 4,7 g Sodium ascorbate - 5,9 g Clear fluids - 1000 ml
  18.00 - 19.00 Clear fluids 500 ml
  19.00 - 20.00 Macrogol-3350 - 100 g Sodium sulfate - 7,5 g Sodium chloride - 2,691 g Potassium chloride - 1,015 g Ascorbic acid - 4,7 g Sodium ascorbate - 5,9 g Clear fluids - 1000 ml
  20.00 - 21.00 Clear fluids 500 ml
  Interventions: Procedure: Mechanical bowel preparation only

INTERVENTIONS:
Procedure: Full bowel preparation — MBP+OA
  Arms: Full bowel preparation (MBP+OA)
Procedure: Mechanical bowel preparation only — MBP
  Arms: Mechanical bowel preparation only

SUMMARY:
The purpose of the study is to determine if short-term outcomes of rectal resections after full bowel preparation (mechanical bowel preparation plus oral antibiotics) are superior to rectal resections with only mechanical bowel preparation.

DETAILED DESCRIPTION:
The design involves random allocation of eligible patients to full bowel preparation or only mechanical bowel preparation in 1:1 ratio. After that rectal resection is performed in both groups.

Short-term outcomes are assessed in 30 day period after surgery. This is a superiority trial evaluating statistical superiority. Rate of surgical site infection is anticipated to decrease from 12% (data from local registry) to 6%. For power of 80% enrolment of 622 patients is required.

The intent-to-treat principle is used for the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the rectum or rectosigmoid junction
* clinical stage T1-4aN0-2M0-1 (distant metastases must be resectable)
* indications for surgical rectal resection
* ECOG status 0-2
* At least 18 years of age
* Written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or comply with the study protocol
* Pregnancy or breast feeding
* Medical contraindications for surgical treatment
* Any use of antibiotics 30 days prior to inclusion
* Functioning stoma
* Contraindications for use of MBP or OA drugs or their components
* Indications for obstructive resection or abdominoperineal excision
* Acute bowel obstruction, bleeding or perforation
* Other malignancies not in remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 622 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Incisional surgical site infection (SSI) rate | 30 days
  Rate of incisional SSI in patients after rectal resections

SECONDARY OUTCOMES:
Anastomotic leak rate | 30 days
  Rate of clinical and/or radiological anastomotic leaks
Intraabdominal and or pelvic abscess rate | 30 days
Overall morbidity | 30 days
  Rate of patients with any complications after surgery
Rate of intraoperative complications | Duration of surgical procedure
Surgery duration in minutes | Duration of surgical procedure
Quality of bowel preparation assessed by surgeon | Day of surgery
  Assessment of bowel preparation quality by surgeon (qualitative scale)
Bowel preparation compliance | Day of surgery
  Rate of patients in experimental arm undergoing complete bowel preparation according to protocol

CONTACTS AND LOCATIONS:
Overall Officials: Aleksei Karachun, Study Chair — National Medical Research Centre of Oncology named after N.N. Petrov
Locations (7):
- Russia (7):
  - GBUZ Moscow Clinical Scientific Center named after Loginov MHD, Moscow
  - I.M. Sechenov First Moscow State Medical University, Clinic of Oncology, Radiotherapy and Reconstructive Surgery, Moscow
  - Lomonosov Moscow State University Medical Research and Educational Center, Moscow
  - Ryazan State Clinical Hospital, Ryazan
  - Scientific-Research institute of Oncology named after N.N. Petrov, Saint Petersburg
  - Tomsk Regional Oncology Hospital, Tomsk
  - Volgograd State Medical University, Ministry of Health of Russia, Volgograd

IPD SHARING:
Plan to Share IPD: No
We are not planning to share individual participant data